CLINICAL TRIAL: NCT03139890
Title: The Effects of Macronutrients on Postprandial Vascular Function in Overweight and Slightly Obese Men
Brief Title: Macronutrients and Postprandial Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 17-3-012
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Dietary Fats; Carbohydrates; Proteins; Macronutrients; Vascular Function; Postprandial Metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-fat milkshake (Experimental)
  Interventions: Other: High-fat (HF-LC-LP) milkshake
- High-carbohydrate milkshake (Experimental)
  Interventions: Other: High-carbohydrate (LF-HC-LP) milkshake
- High-protein milkshake (Experimental)
  Interventions: Other: High-protein (LF-LC-HP) milkshake

INTERVENTIONS:
Other: High-fat (HF-LC-LP) milkshake — During this experimental day, men will receive a high-fat milkshake
  Arms: High-fat milkshake
Other: High-carbohydrate (LF-HC-LP) milkshake — During this experimental day, men will receive a high-carbohydrate milkshake
  Arms: High-carbohydrate milkshake
Other: High-protein (LF-LC-HP) milkshake — During this experimental day, men will receive a high-protein milkshake
  Arms: High-protein milkshake

SUMMARY:
Vascular function decreases following the intake of a mixed meal in some, but not all studies. Differences in the relative amounts of dietary fat, carbohydrates and protein present in the mixed-meal challenges may have contributed to these apparently inconsistent results. Well-designed trials - comparing under rigorously standardized conditions - on the effects of macronutrients on postprandial vascular function are missing. The primary objective of the current study is thus to evaluate in overweight and slightly obese men the effects of the three macronutrients (fat, carbohydrates, and protein) on postprandial vascular function, as assessed by brachial artery flow-mediated vasodilation (FMD). Secondary objectives are to examine postprandial effects on other markers reflecting vascular function, plasma markers for low-grade systemic inflammation and endothelial dysfunction, blood pressure, and serum lipid and plasma glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-70 years
* Men
* BMI between 25-35 kg/m2 (overweight and slightly obese)
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 2.2 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* No current smoker
* No diabetic patients
* No familial hypercholesterolemia
* No abuse of drugs
* No more than 3 alcoholic consumptions per day
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* No use of dietary supplements known to interfere with the main study outcomes as judged by the principal investigator
* No use of medication to treat blood pressure, lipid or glucose metabolism
* No use of an investigational product within another biomedical intervention trial within the previous 1-month
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Women
* Fasting plasma glucose ≥ 7.0 mmol/L
* Fasting serum total cholesterol ≥ 8.0 mmol/L
* Fasting serum triacylglycerol ≥ 2.2 mmol/L
* Systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use of dietary supplements known to interfere with the main study outcomes as judged by the principal investigator
* Use medication to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Not willing to give up being a blood donor from 8 weeks before the start of the study, during the study or for 4 weeks after completion of the study
* Not or difficult to venipuncture as evidenced during the screening visit

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Vascular endothelial function | Change from baseline at 2 hours after milkshake consumption
  Flow-mediated vasodilation (FMD) of the brachial artery

SECONDARY OUTCOMES:
Vascular function markers | Change from baseline at 2 hours after milkshake consumption
  Carotid-femoral pulse wave velocity (PWV), pulse wave analysis (PWA), retinal microvascular caliber
Cardiometabolic risk markers | Change from baseline at 2 hours after milkshake consumption
  Plasma markers for low-grade systemic inflammation and endothelial dysfunction
Cardiometabolic risk markers | During 4 hours following milkshake consumption
  Office blood pressure
Postprandial metabolism | During 4 hours following milkshake consumption
  Serum lipid and plasma glucose metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gravesteijn E, Mensink RP, Smeets ETHC, Plat J. Dietary Macronutrients Do Not Differently Influence Postprandial Serum and Plasma Brain-Derived Neurotrophic Factor Concentrations: A Randomized, Double-Blind, Controlled Cross-Over Trial. Front Neurosci. 2021 Dec 21;15:774915. doi: 10.3389/fnins.2021.774915. eCollection 2021. PMID 34992516
- [Derived] Schroor MM, Plat J, Konings MCJM, Smeets ETHC, Mensink RP. Effect of dietary macronutrients on intestinal cholesterol absorption and endogenous cholesterol synthesis: a randomized crossover trial. Nutr Metab Cardiovasc Dis. 2021 May 6;31(5):1579-1585. doi: 10.1016/j.numecd.2021.01.010. Epub 2021 Jan 29. PMID 33744041
- [Derived] Smeets ETHC, Mensink RP, Joris PJ. Dietary macronutrients do not differently affect postprandial vascular endothelial function in apparently healthy overweight and slightly obese men. Eur J Nutr. 2021 Apr;60(3):1443-1451. doi: 10.1007/s00394-020-02340-y. Epub 2020 Jul 29. PMID 32728881